CLINICAL TRIAL: NCT01567189
Title: Outpatient Cardiac Rehabilitation Versus Hospital. Cost-effectiveness Study
Brief Title: Cost-effectiveness of Outpatient Versus Hospital Cardiac Rehabilitation
Acronym: CERC1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Fernando Arós Borau, Cardiologist, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CERC1
Record Dates: First submitted 2012-02-22; First posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Heart Disease
Keywords: Exercise therapy; cost effectiveness; cardiac rehabilitation; home-based exercise
MeSH Terms: conditions — Coronary Disease | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hospital cardiac rehabilitation (Experimental): The patients will perform physical training sessions in the hospital
  Interventions: Behavioral: Cardiac rehabilitation
- Home cardiac rehabilitation (Active Comparator): The patients will perform physical training sessions at home
  Interventions: Behavioral: Cardiac rehabilitation

INTERVENTIONS:
Behavioral: Cardiac rehabilitation — * Training sessions: 8 weeks of supervised physical training sessions. Stress intensity will be calculated from the peak heart rate reached during stress test: 60-70% during the first month and 70-85% during the second one. Patients will be advised to do at least 1 hour of outdoor exercise with the same intensity on the days when they do not attend hospital.
  * Health education sessions and relaxation sessions: one per week.
  * Smoking and diet checking: as recommended by doctor.
  Arms: Hospital cardiac rehabilitation
Behavioral: Cardiac rehabilitation — The only difference in the hospital's program is that training sessions will be out of hospital with the same target heart rate that in this case will be controlled with pulsometer or Borg scale. The recommended frequency of sessions will be: at least 5 days a week with a minimum of 1 hour / day.
  Arms: Home cardiac rehabilitation

SUMMARY:
The hypothesis is that home based clinical rehabilitation (CR) is less expensive than hospital based CR with similar clinical effectiveness. The investigators will compare the results of two forms of CR on

1. direct and indirect healthcare costs
2. effectiveness on mortality, morbidity, modifiable risk factors control, functional capacity measured by exercise testing, health related quality of life and satisfaction rate
3. cost/effectiveness analysis

DETAILED DESCRIPTION:
The main reasons for patients not to participate in a cardiac rehabilitation program that usually develops by group in the hospital or in a gym, are problems of access to hospital, disgust for participating in a group activity and problems in reconciling their work and / or home with the program schedule. These problems could be overcome by outcome cardiac rehabilitation and thus could increase the number of patients benefit from treatment in either the environment extra or intra-hospital.

Low and medium coronary patients sent to cardiac rehabilitation program at our center within the first 12 weeks after presenting with acute coronary syndrome or been revascularized will be included in the study. The prescription of intensity of effort is based on heart rate reached during the stress test for the initial evaluation in all cases, although at home-program heart rate will be monitored using heart rate monitor and / or by the Borg scale. In this way outpatient group patient could performed training sessions individually and at the time of day that best suits their capabilities. The other program components: control of risk factors, health education and counseling will be identical in both groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* patients referred to cardiac rehabilitation program in the first twelve weeks after an acute coronary syndrome (myocardial infarction or unstable angina) or after percutaneous or surgical revascularization
* who have no contraindication to participate in the program

Exclusion Criteria:

* contraindication to participate in the program
* high-risk criteria for home cardiac rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Morbidity | 1 year
  Readmissions, percutaneous or surgical revascularization
Cost | 1 year
  1. Direct costs
     1. direct healthcare costs: hospital admissions for cardiovascular causes, percutaneous or surgical revascularization, medical and nursing consultation, physical training sessions, medical explorations including the analytic explorations, medication consumption, emergency department visits, depreciation of equipment used.
     2. Direct costs other than health: Transfer the patient for his attention, passenger costs if necessary.
  2. Indirect costs: working days lost during program participation (2 months, family overloads caused by participation in the program (2 months).

SECONDARY OUTCOMES:
Control of risk factors | 1 year
  Control of risk factors at the end of training sessions and one year after the acute event: Percentage of patients achieving the therapeutic goal outlined in the clinical practice guidelines in each of the risk factors
Functional capacity | 1 year
  Oxygen consumption peak measured during exercise testing
Quality of Life | 1 year
  SF-12 version 2
Satisfaction | 1 year
  satisfaction questionnaire based on Osakidetza Basque Health Service questionnaires
Mortality | 1 year
  All cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Araba University Hospital, Vitoria-Gasteiz, Álava, Spain